CLINICAL TRIAL: NCT05740709
Title: Identification of Patients at Risk of Chronic Kidney Disease After Acute Kidney Injury
Brief Title: Identification of Patients at Risk of CKD After AKI
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Guy's and St Thomas' NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: IRAS 319992
Record Dates: First submitted 2022-10-10; First posted 2023-02-23 (Actual); Last update posted 2024-01-23 (Actual); Status verified 2024-01

CONDITIONS: Acute Kidney Injury; Kidney Diseases
Keywords: acute kidney injury; chronic kidney disease; kidney biomarkers
MeSH Terms: conditions — Acute Kidney Injury; Kidney Diseases; Renal Insufficiency, Chronic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — plasma and urine samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- AKI patients: Patients who suffered from AKI whilst in ICU and are awaiting discharge from hospital

SUMMARY:
The investigators will investigate whether new kidney biomarkers can identify patients who are at risk of chronic kidney disease after an episode of moderate / severe acute kidney injury in ICU.

DETAILED DESCRIPTION:
Acute kidney injury (AKI) is a common complication during critical illness and associated with serious short and long-term complications. Participants with AKI have an increased risk of developing dysfunction of other organs, including multi-organ failure, a longer stay in hospital and a higher risk of dying. Survivors remain at risk of complications, even if kidney function initially recovers. In particular, they are at high risk of developing chronic kidney disease, dialysis-dependent end-stage kidney disease and cardiovascular comorbidities. At present, the tools to identify patients at highest risk of chronic kidney disease (CKD) are very limited.

The investigators will recruit participants who had AKI whilst in ICU and are scheduled to be discharged from hospital. Within 3 days of discharge from hospital, blood and urine kidney biomarkers will be measured to explore whether there is a correlation with renal function 3 months later and to identify those at highest risk of CKD. In addition, quality of life at 3 months will be assessed.

ELIGIBILITY:
Inclusion Criteria:

critically ill adult patients who had AKI stage II or III whilst in ICU and are scheduled to be discharged from hospital

Exclusion Criteria:

1. known pre-existing end-stage kidney disease or advanced CKD (stage 3b or worse)
2. kidney transplant within the last 12 months
3. known primary renal disease
4. discharge from hospital for end-of-life care
5. transfer to another health care institution for ongoing in-patient care
6. not expected to survive for 3 months
7. pregnancy
8. lack of capacity to give consent
9. receiving regular dialysis at hospital discharge
10. CKD stage 3 or worse at hospital discharge

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: critically ill adult patients in the ICU
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-03-01 (Actual); Primary Completion 2025-01-01 (Estimated); Study Completion 2026-01-01 (Estimated)

PRIMARY OUTCOMES:
serum creatinine | 3 months after discharge from hospital
  estimated glomerular filtration rate (eGFR) <60ml/min

SECONDARY OUTCOMES:
mortality | 90 days
  mortality
cardiovascular morbidity | 3 months post hospitalisation
  new or worsened cardiovascular morbidity
questionnaire | 3 months post hospitalisation
  health-related quality of life based on questionnaire EQ-5D-5L

CONTACTS AND LOCATIONS:
Overall Officials: Marlies Ostermann, PhD, Principal Investigator — Guy's & St Thomas' NHS Foundation Hospital
Locations (1):
- Guy's & St Thomas Foundation Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No